CLINICAL TRIAL: NCT03614832
Title: Optimal Dose of Ticagrelor（90 mg qd）and Double Standard-dose Clopidogrel on Platelet Aggregation in Clopidogrel Resistance's Patients With Coronary Heart Disease
Brief Title: Ticagrelor and Clopidogrel on Platelet Aggregation in Clopidogrel Resistance's Patients With CHD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHD-201802
Record Dates: First submitted 2018-07-03; First posted 2018-08-03 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-02

CONDITIONS: Platelet Reactivity
Keywords: ticagrelor; clopidogrel; platelet reactivity
MeSH Terms: interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ticagrelor 90 mg (Experimental): To observe low-dose of ticagrelor（90 mg once daily oral）on platelet aggregation in clopidogrel resistance's patients with coronary heart disease.
  Interventions: Drug: Ticagrelor 90 mg
- Clopidogrel 150 mg (Active Comparator): To observe double standard-dose clopidogrel （150 mg once daily oral）on platelet aggregation in clopidogrel resistance's patients with coronary heart disease.
  Interventions: Drug: Clopidogrel 150 mg

INTERVENTIONS:
Drug: Ticagrelor 90 mg — half-dose ticagrelor treatment (90 mg loading dose, then 90 mg once daily) for 1 week.
  Arms: Ticagrelor 90 mg
Drug: Clopidogrel 150 mg — double standard-dose clopidogrel treatment (150 mg loading dose, then 150 mg once daily) for 1 week.
  Arms: Clopidogrel 150 mg

SUMMARY:
The study sought to observe the effects of optimal dose of ticagrelor（90 mg qd）ticagrelor and double standard-dose clopidogrel on platelet reactivity in coronary heart disease patients with high on-treatment platelet reactivity (HTPR) while on clopidogrel.

HTPR with clopidogrel administration in coronary heart disease (CHD) patients has associated with an increased risk of adverse events. Newer P2Y12 inhibitors ticagrelor (90mg BID) provide stronger platelet inhibition compared with clopidogrel, but a low-dose of ticagrelor (90mg QD) has not been previously studied in Chinese CHD patients with HTPR.

DETAILED DESCRIPTION:
Dual antiplatelet therapy (DAPT) with aspirin and P2Y12 receptor inhibitor has been the mainstay for the prevention of recurrent ischemic events in ACS patients and in those undergoing PCI. However, clopidogrel shows major individual variation in its antiplatelet effect in association with an increased incidence of ischemic events and stent thrombosis in patients with High on-treatment platelet reactivity (HTPR). There are several possible mechanisms of clopidogrel response variability or "resistance". Recently, it has been reported that a marked decrease in platelet response to clopidogrel is highly associated with the CYP2C19*2 loss-of-function allele, leading to an adverse prognosis.

Ticagrelor is the first reversibly binding, oral, direct acting P2Y12 receptor antagonist. Increasing studies showed that ticagrelor has a more rapid onset of effect and greater inhibition of platelet aggregation compared with clopidogrel. Recently, it has been reported that low-dose ticagrelor either with 90 mg QD or 45 mg BID, was associated with a more potent antiplatelet effect compared with clopidogrel treatment and once daily dose provided similar antiplatelet effect but favorable effect on optimal platelet inhibition compared with twice daily dose. Hiasa et al. identified that ticagrelor 45 mg twice daily was associated with enhanced inhibition of platelet aggregation (IPA) compared with clopidogrel 75 mg once daily in 118 Japanese patients with stable CAD. In our previous study, the investigators found that half-dose ticagrelor produced similar inhibitory effects on platelet aggregation as standard-dose ticagrelor and exerted significantly stronger effects than clopidogrel in patients with ACS and one-quarter standard-dose ticagrelor provided greater degree of platelet inhibition than clopidogrel in patients with stable CAD. Furthermore, standard-dose ticagrelor (180mg loading dose [LD], then 90mg twice daily) has a significant increase in the risk of bleeding and incidence rate of dyspnea, and that higher discontinuation rates due to adverse effects compared to clopidogrel. A recent study demonstrated that maximum plasma concentration and area under the plasma concentration-time curve of ticagrelor (90 mg twice daily) and its active metabolite (AR-C124910XX) tended to be approximately 40% higher in healthy Chinese volunteers compared with Caucasian subjects. Notably, poor drug metabolism of clopidogrel is more common in Asian populations compared with other international regions, due to the prevalence of CYP2C19 reduced-function alleles. The data suggested that a low dose of ticagrelor might be more appropriate for Chinese patients. Therefore, the optimal dose of ticagrelor for Chinese patients with HTPR is increasingly urgent.

So the objectives of this clinical study were to evaluate the effects of optimal dose of ticagrelor（90 mg qd）ticagrelor and double standard-dose clopidogrel on platelet reactivity in Chinese CHD patients with HTPR.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with coronary heart disease (CHD) ;
2. Patients with high on-treatment platelet reactivity (HTPR) while on clopidogrel. Meet the one standards of the following:

(1) The platelet aggregation rate (PAgR) measured with light transmission aggregometry (LTA) is decreased no more than 10% from baseline level, or PAgR is more than 46%; (2) The percentage of inhibition of ADP-induced platelet aggregation measured by thrombelastogram is not more than 30%; (3) The PRU of inhibition of ADP-induced platelet aggregation measured by VerifyNow >208.

Exclusion Criteria:

1.Severe lung injury; 2.Planned use of glycoprotein IIb/IIIa receptor inhibitors, adenosine diphosphate (ADP) receptor antagonists, or anticoagulant therapy during the study period; 3.Platelet count <100g/L; 4.Creatinine clearance rate < 30ml/min; 5.Severe liver injury. 6.Diagnosed as respiratory or circulatory instability (cardiac shock, severe congestive heart failure NYHA II-IV or left ventricular ejection fraction < 40%); 7.A history of bleeding tendency; 8.Aspirin, ticagrelor or clopidogrel allergies;

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
The plateletinhibition ratio. | up to 7 days
  Thromboelastography (TEG) was used to measure platelet inhibition ratio.

SECONDARY OUTCOMES:
The platelet aggregation ratio. | up to 7 days
  Light transmission aggregometry method was used to measure platelet aggregation

CONTACTS AND LOCATIONS:
Overall Officials: Yue Li, PhD, Principal Investigator — First Affiliated Hospital of Harbin Medical University
Locations (1):
- the first affiliated hospital of Harbin medical university, Harbin, Heilongjiang, China